CLINICAL TRIAL: NCT02711488
Title: Managing Adolescent Obesity at Local Level by Combining Primary and Secondary Intervention
Acronym: PAAPAS-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, MD, PhD. Full Professor of Epidemiology, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMS-PAAPAS-project
Record Dates: First submitted 2016-02-15; First posted 2016-03-17 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: school-based intervention; sedentary behavior; physical activity; sugar sweetened beverages
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Combine primary prevention activities at the school level with secondary prevention at the household level
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Intervention group — The proposed intervention will focus on encouraging students to change their eating habits and food consumption over 9 months (from March to November). Monthly 1-h sessions in the classroom will be given by the class teacher, and includes playing games, staging theater sketches, watching movies and puppet shows, and writing and drawing contests. The activities were designed to discourage students from consuming sugar-sweetened beverages as well as getting them to replace snacks, particularly processed foods (especially cookies) with fresh fruit or healthy homemade food. To reinforce the messages of the in-class nutritional sessions, a set of messages will be sent to the families in the form of illustrated booklets and recipes.
  The secondary prevention strategy at households will be developed for those with excessive weight. The family will receive additional motivation to change these behaviors, using the community health agents as the encourager.
  Arms: Intervention group

SUMMARY:
The objective of the project is to develop, implement and evaluate a prevention program for obesity among adolescents in Brazil combining the primary care health system implemented in the country in recent decades with primary prevention at schools.

DETAILED DESCRIPTION:
The study will combine primary prevention activities at the school level with secondary prevention at the household level, both focusing on behavior strategies such as mindfulness, reduction of eating rate; eating with others at a dinning table; healthy eating, increasing physical activity and reducing sedentary lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

* Both prevention programs
* 5th and 6th grades students
* consent form signed by parents/tutors
* Secondary prevention program
* Overweight and obese children

Exclusion Criteria:

* pregnant girls

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | one year

SECONDARY OUTCOMES:
Body composition | one year
  body composition will be estimated by bioelectrical impedance, using the leg=to=leg method with Tanita scales

OTHER OUTCOMES:
adherence to the protocol at household level | one year
  will be measured by questionnaire
physical activity | one year
  will be measured by questionnaire
physical activity | one year
  In a subgroup will be measured by accelerometer (GT3X Actigraph).
food intake | one year
  Will be assessed by 24-hour recall
food intake | one year
  Will be assessed by a short (23 items) food frequency questionnaire (FFQ), reduced from a validated FFQ for Brazilian adolescents.

REFERENCES:
- [Derived] Sgambato MR, Cunha DB, Henriques VT, Estima CC, Souza BS, Pereira RA, Yokoo EM, Paravidino VB, Sichieri R. PAAPPAS community trial protocol: a randomized study of obesity prevention for adolescents combining school with household intervention. BMC Public Health. 2016 Aug 17;16(1):809. doi: 10.1186/s12889-016-3473-3. PMID 27534742